CLINICAL TRIAL: NCT06223750
Title: Virtual Kidney Check and Follow-up
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Boehringer Ingelheim (Industry); Research Manitoba (Other); Manitoba Health, Seniors and Long-Term Care, Province of Manitoba (Unknown); First Nations Health and Social Secretariat of Manitoba (Unknown); Shared Health Manitoba (Unknown); Seven Oaks General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HS24845 (H2021:170)
Record Dates: First submitted 2023-12-19; First posted 2024-01-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient contact via mail with a letter and laboratory requisition (Other): Patient contact via mail with a letter and laboratory requisition for serum creatinine and urine albumin to creatinine ratio
  Interventions: Other: population-based screening for chronic kidney disease
- Patient and primary care network contact via mail with a letter but no laboratory requisition (Other)
  Interventions: Other: population-based screening for chronic kidney disease

INTERVENTIONS:
Other: population-based screening for chronic kidney disease — Randomized controlled trial that uses an integrated health platform for eligibility and outcome assessments

SUMMARY:
The goal of this clinical trial is to determine the most effective way to complete population-based screening for chronic kidney disease (CKD) in First Nations adults in Manitoba. The main questions it aims to answer are:

* To identify chronic kidney disease in First Nations adults in Manitoba
* To risk stratify patients as low, moderate and high risk of kidney failure and organize active surveillance by risk category
* To initiate treatments to prevent to progression of chronic kidney disease in individuals at risk of kidney failure

Participants will be randomized to:

1. Patient contact via mail with a letter and laboratory requisition for serum creatinine and urine Albumin Creatinine Ratio
2. Patient and primary care network contact via mail with a letter but no laboratory requisition

The primary outcome is the difference between groups in the proportion of individuals who undergo screening for chronic kidney disease within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age>= 18 years
* Resident of Manitoba
* First Nations
* Urban, rural or remote location

Exclusion Criteria:

* Kidney failure (dialysis or transplant)
* chronic kidney disease (estimated Glomerular Filtration Rate <60 milliliter/1.73square meter for 3 months)
* Screening for chronic kidney disease with estimated Glomerular Filtration Rate or Albumin to Creatinine ratio in the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3356 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of individuals who undergo screening for Chronic Kidney Disease (CKD) | 6 months
  The proportion of individuals screened for Chronic Kidney Disease using one screening strategy is compared to the proportion of individuals screened using the other screening strategy.

SECONDARY OUTCOMES:
New diagnosis of CKD (Chronic Kidney Disease) | 5 years
  The proportion of individuals with a new diagnosis of CKD by estimated glomerular filtration rate (eGFR) or albuminuria for each screening strategy
Anti-hyperintensive therapy | 5 years
  The proportion of individuals treated with anti-hyperintensive therapy for each screening strategy
Renin angiotensin aldosterone inhibitor blockade treatment | 5 years
  The proportion of individuals treated with renin angiotensin aldosterone inhibitor blockade for each screening strategy
Sodium Glucose Cotransporter 2 (SGLT2) inhibition treatment | 5 years
  The proportion of individuals treated with Sodium Glucose Cotransporter 2 (SGLT2) inhibition for each screening strategy
Mineral corticoid receptor antagonist treatment | 5 years
  The proportion of individuals treated with a mineral corticoid receptor antagonist for each screening strategy
Statins treatment | 5 years
  The proportion of individuals treated with statins for each screening strategy
Anti-platelet agents treatment | 5 years
  The proportion of individuals treated with anti-platelet agents for each screening strategy
Hospitalizations for diseases | 5 years
  The proportion of individuals treated with hospitalizations for acute coronary syndrome, peripheral vascular disease, cerebrovascular disease or heart failure rate. Urine albumin to creatinine ratio, kidney failure risk equation (KFRE) measurements are also calculated for each screening strategy
The number of antihypertensive medications | 5 years
  The number of antihypertensive medications per individual for each screening strategy
Change in estimated Glomerular Filtration Rate, urine albumin to creatinine ratio, kidney failure risk equation measurements | 5 years
  Change in estimated Glomerular Filtration Rate, urine albumin to creatinine ratio, kidney failure risk equation measurements for each individual
estimated Glomerular Filtration Rate slope | 5 years
  Tracking changes in estimated Glomerular Filtration Rate over time indicates progression of chronic kidney disease for each individual
Number of individuals with 40 % decline in estimated Glomerular Filtration Rate | 5 years
  Number of individuals with 40 % decline in estimated Glomerular Filtration Rate
Number of individuals with kidney failure | 5 years
  Number of individuals with kidney failure
Number of individuals on dialysis | 5 years
  Number of individuals on dialysis
Number of individuals to receive kidney transplant | 5 years
  Number of individuals to receive kidney transplant
Number of individuals who have died | 5 years
  Number of individuals who have died

CONTACTS AND LOCATIONS:
Overall Officials: David Collister, MD, PhD, FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- Chronic Disease Innovation Centre, Winnipeg, Canada